CLINICAL TRIAL: NCT01610128
Title: UCT - Development of an Instrument to Assess Disease Control in Patients With Chronic Urticaria (Urticaria Control Test)
Brief Title: Development of an Urticaria Control Test
Acronym: UCT-D
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, K. Weller, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: UCT-D
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Urticaria
Keywords: urticaria, patient reported outcome
MeSH Terms: conditions — Chronic Urticaria; Urticaria

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic urticaria patients: all patients suffering from chronic types of urticaria (chronic spontaneous urticaria as well as chronic inducible forms such as cold contact urticaria)

SUMMARY:
The aim of the project is to develop a patient reported outcome instrument to assess disease control in chronic urticaria patients (Urticaria Control Test - UCT) of age 12 and older.

ELIGIBILITY:
Inclusion Criteria:

all patients suffering from chronic forms of urticaria are eligible

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients suffering from chronic forms of urticaria
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universitätshautklinik Mainz, Mainz, Rhineland-Palatinate
  - Allergie-Centrum-Charite, Berlin, State of Berlin